CLINICAL TRIAL: NCT04116554
Title: Efficacy of Ultrasound-guided Bilateral Transversus Thoracic Muscle Plane Block as Postoperative Analgesia in Adult Patients Undergoing Open Heart Surgeries: a Randomized Controlled Study.
Brief Title: Bilateral Transversus Thoracic Muscle Plane Block as Analgesic in Open Heart Surgeries by US.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Lecturer of Anesthesiology, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D199
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Analgesia
Keywords: transversus thoracic muscle plane block.; analgesic after open heart surgery.
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (A) (Active Comparator): which will have an ultrasound-guided bilateral transversus thoracic muscle plane (TTP) block by injection of 20 mL of 0.25% bupivacaine and the same procedure will be repeated on the other side.
  Interventions: Drug: 0.25% bupivacaine.
- control group (B) (Sham Comparator): which will have sham block bilaterally by injection of 20 ml of 0.9%saline will be injected on each side.
  Interventions: Device: 0.9%saline

INTERVENTIONS:
Drug: 0.25% bupivacaine. — 20 mL of 0.25% bupivacaine and the same procedure will be repeated on the other side
  Other Names: plain marcaine
  Arms: intervention group (A)
Device: 0.9%saline — 20 ml of 0.9%saline will be injected on each side
  Arms: control group (B)

SUMMARY:
OPEN CARDIAC SURGERY may cause severe postoperative pain and promote a high risk of chronic pain if not treated adequately, that is caused by multiple factors; sternotomy, costotransverse and costovertebral joint distensions, opening of the pericardium, internal mammarian artery harvesting, surgical manipulation of the parietal pleura, chest tube insertion and other musculoskeletal trauma that occurs during surgery.

Adequate analgesia is important not only for patient comfort, but for weaning from ventilator and prevention of respiratory complications. Opioids are used to provide analgesia, but they are associated with significant side effects which include sedation, respiratory depression, nausea, and vomiting.

Severe sternotomy pain in cardiac surgery has been reported in up to 49% of patients at rest and 78% at movement. Of the various options for postoperative pain relief in cardiac surgery, we have chosen an ultrasound-guided transversus thoracic muscle plane (TTP) block versus sham block performed by the anesthesiologist.

Transversus thoracic muscle plane (TTP) block and The pecto-intercostal fascial plane block can block multiple anterior branches of the intercostal nerves (T2 to 6), which dominate the internal mammary region with a single injection bilaterally.

DETAILED DESCRIPTION:
After approval of the institutional ethics committee and written informed consent, (70) patients scheduled for open heart surgery including valve replacement or adult congenital (ASD or VSD) in Fayoum university hospital from May 2019 to November 2020 will be enrolled in this randomized prospective double blinded study.

Patients will be divided into two groups randomized by computer generated random numbers that will be placed in separate opaque envelopes that will be opened by study investigators just before the block.Neither the participants, the study investigators, the attending clinicians, nor the data collectors will be aware of groups' allocation until the study end. The Consolidated Standards of Reporting Trials (CONSORT) recommendations for reporting randomized, controlled clinical trials will be followed.

Group A which will have an ultrasound-guided bilateral transversus thoracic muscle plane (TTP) block.

Group B which will have sham block bilaterally. All patients will be preoperatively examined and investigated by complete blood count, coagulation profile, renal and kidney functions and electrolytes. Electrocardiography, chest x ray and echocardiography will be routinely done. Coronary angiography and carotid arterial duplex will be requested on demand.

Patient will be premedicated by intramuscular injection of 10mg morphine at morning of the operation. Before induction of anesthesia, a five-lead electrocardiography system will be applied to monitor heart rate, rhythm, and ST segments (leads II and V5). A pulse oximeter probe will be attached, and a peripheral venous cannula will be placed. For measurement of arterial pressure and blood sampling, a 20 G cannula will be inserted into either right or left radial artery under local anesthesia. After pre-oxygenation, general anesthesia will be induced by midazolam 2-5 mg, fentanyl (10μg/kg), propofol (3-4mg/Kg), followed by atracurium (0.5 mg/kg).

Trachea will be intubated; patients will be mechanically ventilated with oxygen in air so as to achieve normocarbia. This will be confirmed by radial arterial blood gas analysis and capnogram. An esophageal temperature probe and a Foley catheter will also be placed.

For drug infusion, a triple-lumen central venous catheter will be inserted via the right internal jugular vein.

Anesthesia will be maintained by inhaled Isoflurane 0.4 to 1% and atracurium infusion at a rate of 0.5 mg/kg/h for continued muscle relaxation. During extracorporeal circulation, patients will receive propofol infusion at a rate of 50-100 µ/kg/min. in addition to atracurium infusion.

Before initiation of cardiopulmonary bypass (CPB), the patients will receive intravenous heparin (300-500 units/kg body weight) to achieve an activated clotting time >480s. CPB will be instituted via an ascending aortic cannula and a two-stage right atrial cannula. Before, during (pump blood flow: 2.4l/min/m2), and after CPB, mean arterial pressure will be adjusted to exceed 60mmHg. Cardiac arrest will be induced with cold ante-grade blood cardioplegia. Lactate-enriched Ringer's solution will be added to the CPB circuit to maintain reservoir volume when needed, and packed red blood cells will be added when hemoglobin concentration decrease to less than 7g/dl.

After rewarming the patient to 37°C and separation from CPB; reversal of heparin by protamine sulfate (1:1), and sternal closure will be achieved. The study solution (bupivacaine 0.25% or normal saline will be prepared in the operating room by anesthesiology intern). For carrying out either block bilaterally the skin on either side of the sternum will be prepared with povidone iodine solution. Then a linear ultrasound probe (Philips clear vue350, Philips healthcare, Andover MAO1810, USA, Machine ID: 1385, Nile medical center, service@nilemed.net) will be placed on the right and left sides at 3cm from the midsternum. On the surface plane, the subcutaneous tissue is identified, in the intermediate plane, the pectoralis major muscle, the intercostal muscles and the ribs, and in the deep plane the transverse thoracic muscle, the pleura and the lungs.

Group A: will have an ultrasound-guided bilateral transversus thoracic muscle plane (TTP) block. After identification of the anatomical plane between the internal intercostal and the transversus thoracic muscles a 22-gauge short bevel needle (Spinocan, B. Braun Melsungen AG, Germany) will be inserted between the fourth and fifth ribs connecting at the sternum.

Correct needle placement will be confirmed by visualizing the needle in plane along its entire length and the tip of the needle between both muscles, then1 ml of anesthetic liquid will be introduced after confirming a negative aspiration. Appropriate injection to accomplish the TTP block will be indicated by Local anesthetic spread deep to the costal cartilages and downward displacement of the pleura. The TTP blocks will be administered by injection of 20 mL of 0.25% bupivacaine and the same procedure will be repeated on the other side.

Group B: will have sham block bilaterally. The same technique of TTP block will be used to do sham block on either sides of the chest. 20 ml of 0.9%saline will be injected on each side.

Tracheal extubation will be performed when the patient met the following criteria: awake/arousable, hemodynamically stable, no active bleeding, warm peripheries, and satisfactory arterial blood gas with an FIO2 < 0.5, pressure support on ventilator reduced to 10 Cm H2O, Positive End Expiratory Pressure 5-7 CmH2O, no electrolyte abnormalities, minimal inotropic support, or no escalation in inotropic support.

Postoperative analgesia in ICU will be carried out for both groups with the conventional way by the intensivest using opioids (fentanyl), and the total 24 h. opioid consumption will be recorded.

Measured parameters:

The primary outcome is Total opioid (fentanyl) consumption (time frame: from the time of ICU admission up to 24 h).

Secondary outcomes will include:

1. VAS score for sternal pain both during rest and with cough (ranging from 0 indicating no pain to 10 indicating extreme pain) judged by objective pain score (table: 1) measured at time intervals: 30 minutes, 1h., 3h.,6h.,12h., and 24h.
2. Time to extubation (time frame: from the time of ICU admission up to 24 h).
3. Patient satisfaction (measured as poor, good or excellent).
4. Hemodynamic variables (HR, SaO2, MABP and inotropic support). (Time frame: from the time of ICU admission up to 24 h).
5. Nausea and vomiting.
6. Other complications including; infection, hematoma or local anesthetic toxicity.
7. ICU length of stay (Time frame: from the time of ICU admission up to discharge to the ward).
8. Total length stay of hospital (in days).

STATISTICAL ANALYSIS AND SAMPLE SIZE ESTIMATION:

Sample size was calculated using (G power version 3). Minimal sample size of patients was 31 in each group needed to get power level 0.90, alpha level 0.05 and 30% as a difference between the two groups in the morphine consumption after the intervention. To overcome problem of loss of follow up, calculated sample size was increased by 10% to reach 35 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older (18 - 80 yrs. old).
* Scheduled for elective cardiac surgery for valve replacement or adult congenital (VSD or ASD) via median sternotomy.

Exclusion Criteria:

* Patients with emergency surgeries.
* Allergy to drug used.
* re-do surgery.
* Coagulopathy.
* Neuromuscular disease.
* Preoperative poor left ventricular function (EF < 35%).
* Systemic infections or infections at site of injection.
* Psychiatric illnesses (schizophrenia, bipolar, uncontrolled anxiety or depression).
* Narcotic dependency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | from the time of ICU admission hour 1 up to 24 hour
  the amount of opioid (mostly used is fentanyl amp. in equivalent doses ) that has been used for 24 hours after admission in ICU

CONTACTS AND LOCATIONS:
Overall Officials: mohamed hamed, MD, Principal Investigator — Fayoum University; Mahdy ahmed, MD, Principal Investigator — Fayoum University
Locations (1):
- Fayoum University Hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bignami E, Castella A, Allegri M. Postoperative Pain After Cardiac Surgery: An Open Issue. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):e24-e25. doi: 10.1053/j.jvca.2017.09.022. Epub 2017 Sep 20. No abstract available. PMID 29217242
- [Background] Landoni G, Isella F, Greco M, Zangrillo A, Royse CF. Benefits and risks of epidural analgesia in cardiac surgery. Br J Anaesth. 2015 Jul;115(1):25-32. doi: 10.1093/bja/aev201. PMID 26089444
- [Background] Lahtinen P, Kokki H, Hynynen M. Pain after cardiac surgery: a prospective cohort study of 1-year incidence and intensity. Anesthesiology. 2006 Oct;105(4):794-800. doi: 10.1097/00000542-200610000-00026. PMID 17006079